CLINICAL TRIAL: NCT00858767
Title: Comparison of Absorption and Efficacy of 3 Different Menaquinone-7 Delivery Systems; Casein Powder, Arabic Gum Powder, or Linseed Oil
Brief Title: Arabic Gum-Absorption Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Dr. C. Vermeer, VitaK BV
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-3-064
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Bioavailability
Keywords: vitamin K2; absorption; efficacy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 2 casein capsules per day existing of 90 µg menaquinone-7 per day for 8 weeks
  Interventions: Dietary Supplement: menaquinone-7 from casein capsules
- 2 (Active Comparator): 2 arabic gum capsules per day existing of 90 µg menaquinone-7 per day for 8 weeks
  Interventions: Dietary Supplement: menaquinone-7 from arabic gum capsules
- 3 (Active Comparator): 2 linseed capsules existing of 90 µg menaquinone-7 per day for 8 weeks
  Interventions: Dietary Supplement: menaquinone-7 from linseed oil capsules

INTERVENTIONS:
Dietary Supplement: menaquinone-7 from casein capsules — 90 µg menaquinone-7 daily during 8 weeks
  Arms: 1
Dietary Supplement: menaquinone-7 from arabic gum capsules — 90 µg menaquinone-7 daily during 8 weeks
  Arms: 2
Dietary Supplement: menaquinone-7 from linseed oil capsules — 90 µg menaquinone-7 daily during 8 weeks
  Arms: 3

SUMMARY:
Previous studies have indicated that menaquinone-7 (MK-7) is the most effective form of vitamin K. The Japanese soya product natto is one of the richest food sources of MK-7, but its taste is not appreciated by the Western society. For this reason, the active biological compound has been manufactured as enriched oil or casein (≈80% of proteins in cow's milk)-enriched powder. However, cow's milk allergy is the most common cause of food allergy affecting a minimum of 2-3% of infants. The investigators will therefore compare this protein-delivery system to an alternative delivery system (Arabic gum; 98% polysaccharides). To compare the difference between powder and oil as MK-7 delivery vehicle, the investigators will also test the efficacy of enriched linseed oil.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged between 20 and 40 y
* Normal body weight and height (BMI <30 kg/m2)
* Stable body weight (weight gain or loss <3 kg in past 3 mo)
* Caucasian race
* Written consent to take part in the study
* Low vitamin K status

Exclusion Criteria:

* (A history of) metabolic or gastrointestinal diseases
* Chronic degenerative and/or inflammatory diseases
* Abuse of drugs and/or alcohol
* Use of corticosteroids
* Use of oral anticoagulants
* (A history of) soy allergy
* Use of vitamin K-containing multivitamins or vitamin K supplements
* Anaemia
* Blood donation or participation in another study within one month before the study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
serum level menaquinone-7 | 8 weeks

SECONDARY OUTCOMES:
plasma level of biochemical markers carboxylated matrix-Gla protein, undercarboxylated matrix-Gla protein, carboxylated osteocalcin, undercarboxylated osteocalcin | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — VitaK /University of Maastricht
Locations (1):
- VitaK BV /University of Maastricht, Maastricht, Netherlands